CLINICAL TRIAL: NCT03707977
Title: A Clinical Trial to Evaluate the Impact of Broadly Neutralizing Antibodies VRC01LS and 10-1074 on Maintenance of HIV Suppression in a Cohort of Early-Treated Children in Botswana (Dual bNAb Treatment in Children)
Brief Title: Dual bNAb Treatment in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tatelo Study; 38551 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2023-01

CONDITIONS: HIV Infection
Keywords: broadly neutralizing antibodies; HIV suppression
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group PK-A: ART + VRC01LS (Experimental): In the PK Step, participants will continue ART and receive VRC01LS at Weeks 0, 4, and 8 as a single intravenous (IV) dose (30 mg/kg load then 10 mg/kg maintenance).
  Interventions: Drug: ART; Biological: VRC01LS
- Group PK-B: ART + 10-1074 (Experimental): In the PK Step, participants will continue ART and receive 10-1074 at Weeks 0, 4, and 8 as a single IV dose (30 mg/kg).
  Interventions: Drug: ART; Biological: 10-1074
- Steps 1-3 Participants (ART + 10-1074 + VRC01LS) (Experimental): In Step 1, eligible participants will continue to receive ART and will receive both 10-1074 and VRC01LS at Weeks 0, 4, and 8. Following a recommendation from the study team and Safety Monitoring Committee (SMC) to increase the maintenance dosing based on the PK Step, a VRC01LS loading dose of 30 mg/kg will be given at the start of Step 1, followed by 15 mg/kg dosing at each 4-weekly visit, and 10-1074 dosing will be at 30 mg/kg at each 4-weekly visit. In Step 2, participants with ongoing viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks. In Step 3, both 10-1074 and VRC01LS will be discontinued and ART will be re-started.
  Interventions: Drug: ART; Biological: VRC01LS; Biological: 10-1074

INTERVENTIONS:
Drug: ART — ART will not be provided by the study. Participants will continue to receive their ART regimen they were receiving prior to enrolling in the study.
Biological: VRC01LS — Administered by intravenous (IV) infusion
  Arms: Group PK-A: ART + VRC01LS; Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Biological: 10-1074 — Administered by intravenous (IV) infusion
  Arms: Group PK-B: ART + 10-1074; Steps 1-3 Participants (ART + 10-1074 + VRC01LS)

SUMMARY:
The purpose of this study is to evaluate the impact of two broadly neutralizing antibodies, VRC01LS and 10-1074, on the maintenance of HIV suppression in a cohort of early-treated children in Botswana.

DETAILED DESCRIPTION:
This study will evaluate the impact of two broadly neutralizing antibodies, VRC01LS and 10-1074, on the maintenance of HIV suppression in a cohort of early-treated children in Botswana.

The primary objectives are as follows:

1. To conduct an interventional clinical trial to determine the safety, pharmacokinetics, dosing and antiviral efficacy of up to 24 weeks of maintenance VRC01LS and 10-1074 immunotherapy in early-treated HIV-1 infected children in Botswana.
2. To evaluate effects of treatment with VRC01LS and 10-1074 on the size and cellular composition of residual viral reservoirs.
3. To investigate the influence of VRC01LS and 10-1074 treatment on the magnitude and quality of antiviral innate and adaptive immune responses.

The study includes 4 steps: the pharmacokinetics (PK) Step, Step 1, Step 2, and Step 3. In the PK Step, antiretroviral treatment (ART) is continued and 12 study participants will undergo safety and PK testing, 6 for each bNAb used in the study (10-1074 and VRC01LS). In Step 1, ART is continued and dual bNAb treatment occurs, with PK confirmation of dual bNAb dosing for the first 6 participants in Step 1. In Step 2, ART is withdrawn and dual bNAb maintenance treatment occurs. In Step 3, dual bNAbs will be discontinued and participants will be re-started on ART.

Participants will be in the study for a minimum of 56 weeks, and a maximum of 98 weeks for those who start in the PK step and continue through the study.

ELIGIBILITY:
Inclusion Criteria for PK Step*:

* On ART for at least 96 weeks
* Greater than or equal to 96 weeks and less than 5 years of age at enrollment
* HIV RNA less than 40 copies/mL for at least 24 weeks prior to entry
* Ability to remain in close study follow-up for at least 12 weeks
* Willingness to receive IV infusions of bNAbs
* Willingness to provide signed informed consent (by the parent/guardian)

  * *It is anticipated that all children in PK Step will be from Early Infant Treatment (EIT) Study (NCT02369406); however, up to 4 HIV+ children outside the PK Study (age range 2-5 years) may participate in the PK Step if otherwise eligible and if EIT children are unavailable.

Inclusion Criteria for Entry into Step 1 (followed by participation in Steps 2-3):

* EIT Study participant (NCT02369406)
* On ART for at least 96 weeks
* Greater than or equal to 96 weeks and less than 7 years of age at enrollment
* HIV RNA less than 40 copies/mL for at least 24 weeks prior to entry
* Ability to remain in close study follow-up for at least 56 weeks
* Willingness to receive IV infusions of bNAbs
* Willingness to provide signed informed consent (by the parent/guardian)

Exclusion Criteria:

* Medical condition making survival for at least 32 weeks unlikely
* Active tuberculosis or malignancy
* Actively breastfeeding
* Previous receipt of VRC01/VRC01LS or 10-1074 (except during the PK Step)

Ages: 96 Weeks to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Shapiro, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH); Daniel Kuritzkes, MD, Principal Investigator — Brigham and Women's Hospital; Mathias Lichterfeld, MD, PhD, Principal Investigator — Brigham and Women's Hospital/Massachusetts General Hospital
Locations (2):
- Botswana (2):
  - Francistown Non-Network CRS, Francistown
  - Botswana Harvard AIDS Institute Partnership CRS Non-Network, Gaborone

REFERENCES:
- [Result] Capparelli EV, Ajibola G, Maswabi K, Holme MP, Bennett K, Powis KM, Moyo S, Mohammed T, Maphorisa C, Hughes MD, Seaton KE, Tomaras GD, Mosher S, Taylor A, O'Connell S, Narpala S, Mcdermott A, Caskey M, Gama L, Lockman S, Jean-Philippe P, Makhema J, Kuritzkes DR, Lichterfeld M, Shapiro RL; Tatelo Study Team. Safety and Pharmacokinetics of Intravenous 10-1074 and VRC01LS in Young Children. J Acquir Immune Defic Syndr. 2022 Oct 1;91(2):182-188. doi: 10.1097/QAI.0000000000003033. PMID 36094485
- [Result] Shapiro RL, Ajibola G, Maswabi K, Hughes M, Nelson BS, Niesar A, Pretorius Holme M, Powis KM, Sakoi M, Batlang O, Moyo S, Mohammed T, Maphorisa C, Bennett K, Hu Z, Giguel F, Reeves JD, Reeves MA, Gao C, Yu X, Ackerman ME, McDermott A, Cooper M, Caskey M, Gama L, Jean-Philippe P, Yin DE, Capparelli EV, Lockman S, Makhema J, Kuritzkes DR, Lichterfeld M. Broadly neutralizing antibody treatment maintained HIV suppression in children with favorable reservoir characteristics in Botswana. Sci Transl Med. 2023 Jul 5;15(703):eadh0004. doi: 10.1126/scitranslmed.adh0004. Epub 2023 Jul 5. PMID 37406137
- [Result] Banga J, Nelson BS, Ajibola G, Mohammed T, Maphorisa C, Boleo C, Moyo S, Batlang O, Sakoi-Mosetlhi M, Maswabi K, Holme MP, Powis KM, Lockman S, Hughes MD, Makhema J, Kuritzkes DR, Litcherfeld M, Shapiro R. Predictive markers for sustained viral suppression on dual bNAbs during ART interruption in children. J Acquir Immune Defic Syndr. 2025 Mar 26:10.1097/QAI.0000000000003663. doi: 10.1097/QAI.0000000000003663. Online ahead of print. PMID 40136003
- [Result] Sakoi-Mosetlhi M, Ajibola G, Haghighat R, Batlang O, Maswabi K, Pretorius-Holme M, Powis KM, Lockman S, Makhema J, Litcherfeld M, Kuritzkes DR, Shapiro R. Caregivers of children with HIV in Botswana prefer monthly IV Broadly Neutralizing Antibodies (bNAbs) to daily oral ART. PLoS One. 2024 Mar 27;19(3):e0299942. doi: 10.1371/journal.pone.0299942. eCollection 2024. PMID 38536810

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PK Step was a lead-in to the main study. Twelve participants enrolled in and completed the PK Step (Group PK-A or Group PK-B). Ten of the 12 participants from the PK Groups later enrolled in Step 1, and 18 additional participants who had not participated in the PK Step enrolled in Step 1 for a total of 28 participants to enter Step 1 (and then progress to Step 2 and/or Step 3). Thirty participants enrolled overall in the PK Step and/or the main study.
Groups:
- Steps 1-3 Participants (ART + 10-1074 + VRC01LS, Then 10-1074 + VRC01LS Only, Then ART Only): In Step 1, eligible participants will continue to receive ART and will receive both 10-1074 and VRC01LS at Weeks 0, 4, and 8. Following a recommendation from the study team and Safety Monitoring Committee (SMC) to increase the maintenance dosing based on the PK Step, a VRC01LS loading dose of 30 mg/kg will be given at the start of Step 1, followed by 15 mg/kg dosing at each 4-weekly visit, and 10-1074 dosing will be at 30 mg/kg at each 4-weekly visit.
  In Step 2, participants with ongoing viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks.
  In Step 3, both 10-1074 and VRC01LS will be discontinued and ART will be re-started.
  ART: ART will not be provided by the study. Participants will continue to receive their ART regimen they were receiving prior to enrolling in the study.
  VRC01LS: Administered by intravenous (IV) infusion
  10-1074: Administered by intravenous (IV) infusion
Period: PK Step
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS, Then 10-1074 + VRC01LS Only, Then ART Only)
Started | 6 | 6 | 0
Completed | 6 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Steps 1 (ART+bNAbs)
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS, Then 10-1074 + VRC01LS Only, Then ART Only)
Started | 0 | 0 | 28
Completed | 0 | 0 | 25
Not Completed | 0 | 0 | 3
Not completed — HIV-1 RNA >40 copies/mL while receiving ART + bNAbs in Step 1 | 0 | 0 | 3
Period: Step 2 (bNAbs Only)
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS, Then 10-1074 + VRC01LS Only, Then ART Only)
Started | 0 | 0 | 25
Completed | 0 | 0 | 11
Not Completed | 0 | 0 | 14
Not completed — HIV-1 RNA >400 copies/mL while receiving bNAbs alone in Step 2 | 0 | 0 | 14
Period: Step 3 (Stop bNABs, Resume ART)
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS, Then 10-1074 + VRC01LS Only, Then ART Only)
Started | 0 | 0 | 28
Completed | 0 | 0 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants who entered the PK Step (a lead-in to the main study) in Group B did not proceed to Step 1 due to ineligibility for Step 1. Baseline characteristics of these 2 participants are reported separately. Baseline characteristics (at the time of study entry) for all 28 other participants (including those who entered the study in the PK Step and proceeded to Step 1) are shown in the Steps 1-3 group results.
Groups:
- Steps 1-3 Participants (ART + 10-1074 + VRC01LS): In Step 1, eligible participants will continue to receive ART and will receive both 10-1074 and VRC01LS at Weeks 0, 4, and 8. A VRC01LS loading dose of 30 mg/kg will be given at the start of Step 1, followed by 15 mg/kg dosing at each 4-weekly visit, and 10-1074 dosing will be at 30 mg/kg at each 4-weekly visit. In Step 2, participants with ongoing viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks. In Step 3, both 10-1074 and VRC01LS will be discontinued and ART will be re-started.
- Total: Total of all reporting groups
Arm/Group | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS) | Total
Number analyzed (Participants) | 2 | 28 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at study entry
  years | 3.12 [2.13 to 4.10] | 3.29 [2.80 to 3.98] | 3.29 [2.70 to 4.10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 19 | 21
  Male | 0 | 9 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Botswana | 2 | 28 | 30
Weight [Median (Inter-Quartile Range); unit: kg] — Weight at study entry
  kg | 12.85 [10.30 to 15.40] | 12.55 [11.00 to 14.65] | 12.55 [10.90 to 15.20]
Height [Median (Inter-Quartile Range); unit: cm] — Height at study entry
  cm | 94 [85 to 103] | 94 [87.5 to 101.5] | 94 [87 to 102]
CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — CD4 cell count at study entry
  cells/mm^3 | 1173 [1131 to 1215] | 1106 [795 to 1539] | 1124 [833 to 1408]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment-associated Adverse Events (AEs) [Number of Participants With Treatment-associated Adverse Event(s) of Any Grade]
Time Frame: Measured until 30 days after study completion for each participant
Measure: Count of Participants; unit: Participants
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 6 | 6 | 28
Participants | 4 | 1 | 19

2. Primary Outcome: Severity of Treatment-associated AEs (Number of Participants With Grade 3 or Higher Related AEs)
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table). The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with Grade 1 indicating a mild event, Grade 2 indicating a moderate event, Grade 3 indicating a severe event, Grade 4 indicating a potentially life-threatening event, and Grade 5 indicating death.
Time Frame: Measured until 30 days after study completion for each participant
Measure: Count of Participants; unit: Participants
Groups:
- Group PK-B: ART + 10-1074: n the PK Step, participants will continue ART and receive 10-1074 at Weeks 0, 4, and 8 as a single IV dose (30 mg/kg).
  ART: ART will not be provided by the study. Participants will continue to receive their ART regimen they were receiving prior to enrolling in the study.
  10-1074: Administered by intravenous (IV) infusion
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074 | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 6 | 6 | 28
Participants
  Number of participants with Grade 3 treatment-associated AEs | 0 | 0 | 1
  Number of participants with Grade 4 treatment-associated AEs | 0 | 0 | 0
  Number of participants with Grade 5 treatment-associated AEs | 0 | 0 | 0

3. Primary Outcome: Proportion of Children Who Maintain HIV-1 Plasma RNA Less Than 400 Copies/mL, After Initiating VRC01LS and 10-1074 Infusions and Stopping ART
Description: Based on laboratory evaluations
Time Frame: Measured through Week 24 of Step 2
Measure: Count of Participants; unit: Participants
Groups:
- Steps 2 Participants (10-1074 + VRC01LS): In Step 2, participants who had viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks.
Arm/Group | Steps 2 Participants (10-1074 + VRC01LS)
Number analyzed (Participants) | 25
Participants | 11

4. Primary Outcome: Proportion of Children Who Maintain HIV-1 Plasma RNA Less Than 40 Copies/mL, After Initiating VRC01LS and 10-1074 Infusions and Stopping ART
Description: Based on laboratory evaluations
Time Frame: Measured through Week 24 of Step 2
Measure: Count of Participants; unit: Participants
Groups:
- Steps 2 Participants (10-1074 + VRC01LS): In Step 2, participants who had ongoing viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks.
Arm/Group | Steps 2 Participants (10-1074 + VRC01LS)
Number analyzed (Participants) | 25
Participants | 10

5. Secondary Outcome: VRC01LS or 10-1074 Concentrations in Plasma
Description: Median pre-dose trough (28 days post previous dose) based on laboratory evaluations
Time Frame: Measured through Week 12 (PK Step)
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074
Number analyzed (Participants) | 6 | 6
mcg/mL
  Day 28 | 223.3 [157.9 to 253.3] | 155.2 [91.3 to 318.6]
  Day 56 | 180.7 [164.9 to 227.1] | 232.0 [113.6 to 328.5]
  Day 84 | 156.9 [125.8 to 201.4] | 258.3 [122.4 to 467.3]

6. Secondary Outcome: Median Trough Concentration of VRC01LS or 10-1074 in Plasma 28 Days After the Third Dose
Description: Based on laboratory evaluations
Time Frame: Measured through Week 12 (PK Step)
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Group PK-A: ART + VRC01LS | Group PK-B: ART + 10-1074
Number analyzed (Participants) | 6 | 6
mcg/mL | 156.9 [125.8 to 201.4] | 258.3 [122.4 to 467.3]

7. Secondary Outcome: VRC01LS and 10-1074 Concentrations in Plasma for Each Time Point
Description: Based on laboratory evaluations
Time Frame: Measured through Week 32 following Step 1 entry
Population: The first 6 participants to enter Step 1 were included in a PK analysis to confirm targets were met with dual bNAb administration. Only these 6 participants had PK measurements at Step 1 Week 8. Twenty-five participants in total contributed PK data but those who discontinued bNAbs early due to HIV-1 RNA >400 copies/mL had fewer PK measurements.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 25
mcg/mL
  Step 1 Week 4 (10-1074) | 154.4 [83.7 to 257.2]
  Step 1 Week 8 (10-1074): number analyzed (Participants) | 6
  Step 1 Week 8 (10-1074) | 168.1 [95.5 to 264.7]
  Step 2 Week 0 (10-1074) | 194.6 [120.1 to 417.7]
  Step 2 Week 4 (10-1074): number analyzed (Participants) | 20
  Step 2 Week 4 (10-1074) | 205.6 [125.3 to 404]
  Step 2 Week 8 (10-1074): number analyzed (Participants) | 16
  Step 2 Week 8 (10-1074) | 232.3 [120.3 to 323.2]
  Step 2 Week 12 (10-1074): number analyzed (Participants) | 14
  Step 2 Week 12 (10-1074) | 211.7 [111.2 to 371.5]
  Step 2 Week 16 (10-1074): number analyzed (Participants) | 13
  Step 2 Week 16 (10-1074) | 212.5 [183.6 to 381.6]
  Step 2 Week 20 (10-1074): number analyzed (Participants) | 13
  Step 2 Week 20 (10-1074) | 246.8 [163.5 to 345.8]
  Step 2 Week 24 or Step 3 Entry (10-1074): number analyzed (Participants) | 24
  Step 2 Week 24 or Step 3 Entry (10-1074) | 268.1 [108.5 to 1724.1]
  Step 1 Week 4 (VRC01LS): number analyzed (Participants) | 24
  Step 1 Week 4 (VRC01LS) | 226.5 [139 to 426.3]
  Step 1 Week 8 (VRC01LS): number analyzed (Participants) | 6
  Step 1 Week 8 (VRC01LS) | 293.4 [208 to 329.9]
  Step 2 Week 0 (VRC01LS) | 239.1 [142.7 to 377.4]
  Step 2 Week 4 (VRC01LS): number analyzed (Participants) | 20
  Step 2 Week 4 (VRC01LS) | 255.9 [124.8 to 370.7]
  Step 2 Week 8 (VRC01LS): number analyzed (Participants) | 16
  Step 2 Week 8 (VRC01LS) | 254.7 [104.7 to 497.8]
  Step 2 Week 12 (VRC01LS): number analyzed (Participants) | 14
  Step 2 Week 12 (VRC01LS) | 260.2 [141.8 to 595.3]
  Step 2 Week 16 (VRC01LS): number analyzed (Participants) | 13
  Step 2 Week 16 (VRC01LS) | 273.9 [141.2 to 673.2]
  Step 2 Week 20 (VRC01LS): number analyzed (Participants) | 13
  Step 2 Week 20 (VRC01LS) | 266.5 [154.2 to 663.9]
  Step 2 Week 24 or Step 3 Entry (VRC01LS): number analyzed (Participants) | 24
  Step 2 Week 24 or Step 3 Entry (VRC01LS) | 295.3 [170.9 to 507.8]

8. Secondary Outcome: Proportion of Children With Trough VRC01LS and 10-1074 Concentrations Below Defined Trough Ranges
Description: Based on laboratory evaluations
Time Frame: Measured through Week 32 following Step 1 entry
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 25
Participants
  Step 1 Week 4 (10-1074) | 0
  Step 1 Week 8 (10-1074): number analyzed (Participants) | 6
  Step 1 Week 8 (10-1074) | 0
  Step 2 Week 0 (10-1074) | 0
  Step 2 Week 4 (10-1074): number analyzed (Participants) | 20
  Step 2 Week 4 (10-1074) | 0
  Step 2 Week 8 (10-1074): number analyzed (Participants) | 16
  Step 2 Week 8 (10-1074) | 0
  Step 2 Week 12 (10-1074): number analyzed (Participants) | 14
  Step 2 Week 12 (10-1074) | 0
  Step 2 Week 16 (10-1074): number analyzed (Participants) | 13
  Step 2 Week 16 (10-1074) | 0
  Step 2 Week 20 (10-1074): number analyzed (Participants) | 13
  Step 2 Week 20 (10-1074) | 0
  Step 2 Week 24 or Step 3 entry (10-1074): number analyzed (Participants) | 24
  Step 2 Week 24 or Step 3 entry (10-1074) | 0
  Step 1 Week 4 (VRC01LS): number analyzed (Participants) | 24
  Step 1 Week 4 (VRC01LS) | 2
  Step 1 Week 8 (VRC01LS): number analyzed (Participants) | 6
  Step 1 Week 8 (VRC01LS) | 0
  Step 2 Week 0 (VRC01LS) | 4
  Step 2 Week 4 (VRC01LS): number analyzed (Participants) | 20
  Step 2 Week 4 (VRC01LS) | 1
  Step 2 Week 8 (VRC01LS): number analyzed (Participants) | 16
  Step 2 Week 8 (VRC01LS) | 2
  Step 2 Week 12 (VRC01LS): number analyzed (Participants) | 14
  Step 2 Week 12 (VRC01LS) | 2
  Step 2 Week 16 (VRC01LS): number analyzed (Participants) | 13
  Step 2 Week 16 (VRC01LS) | 1
  Step 2 Week 20 (VRC01LS): number analyzed (Participants) | 13
  Step 2 Week 20 (VRC01LS) | 1
  Step 2 Week 24 or Step 3 entry (VRC01LS): number analyzed (Participants) | 24
  Step 2 Week 24 or Step 3 entry (VRC01LS) | 0

9. Secondary Outcome: Height Z-scores of Virally Suppressed Children Receiving bNAbs
Description: World Health Organization (WHO) standardized Z-scores will be evaluated for changes over time: WHO Length/height-for-age z-score (0-19 yrs), Change from Step 1, Day 0 to Step 3, Week 24. A z-score of 0 corresponds to the population mean. Scores above 0 indicate a participant's height is above the mean, while a score below 0 indicates a participant's height is below the mean. A positive change in z-score corresponds to a higher z-score at the second timepoint compared to the first.
Time Frame: Measured through Week 24 (Step 3)
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 28
change in score on a scale | 0.18 [0.07 to 0.30]

10. Secondary Outcome: Weight Z-scores of Virally Suppressed Children Receiving bNAbs
Description: WHO standardized Z-scores will be evaluated for changes over time: WHO Weight-for-age z-score (0-10 yrs), Change from Step 1, Day 0 to Step 3, Week 24. A z-score of 0 corresponds to the population mean. Scores above 0 indicate a participant's weight is above the mean, while a score below 0 indicates a participant's weight is below the mean. A positive change in z-score corresponds to a higher z-score at the second timepoint compared to the first.
Time Frame: Measured through Week 24 (Step 3)
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | Steps 1-3 Participants (ART + 10-1074 + VRC01LS)
Number analyzed (Participants) | 28
change in score on a scale | 0.09 [0.04 to 0.22]

ADVERSE EVENTS:
Time Frame: Measured until 30 days after study completion for each participant. Each column reports events occurring during that specific step.
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)
Groups:
- PK Step (ART + VRC01LS): In the PK Step, participants will continue ART and receive VRC01LS at Weeks 0, 4, and 8 as a single intravenous (IV) dose (30 mg/kg load then 10 mg/kg maintenance).
  ART: ART will not be provided by the study. Participants will continue to receive their ART regimen they were receiving prior to enrolling in the study.
  VRC01LS: Administered by intravenous (IV) infusion
- PK Step (ART + 10-1074): In the PK Step, participants will continue ART and receive 10-1074 at Weeks 0, 4, and 8 as a single IV dose (30 mg/kg).
  ART: ART will not be provided by the study. Participants will continue to receive their ART regimen they were receiving prior to enrolling in the study.
  10-1074: Administered by intravenous (IV) infusion
- Step 1 (ART + VRC01LS + 10-1074): In Step 1, eligible participants will continue to receive ART and will receive both 10-1074 and VRC01LS at Weeks 0, 4, and 8. A VRC01LS loading dose of 30 mg/kg will be given at the start of Step 1, followed by 15 mg/kg dosing at each 4-weekly visit, and 10-1074 dosing will be at 30 mg/kg at each 4-weekly visit.
- Step 2 (VRC01LS + 10-1074 Only): In Step 2, participants with ongoing viral suppression throughout Step 1 will undergo withdrawal of ART and will continue maintenance 10-1074 (30 mg/kg) and VRC01LS (15 mg/kg) treatment for up to 24 weeks.
- Step 3 (ART Only): In Step 3, both 10-1074 and VRC01LS will be discontinued and ART will be re-started.
Arm/Group | PK Step (ART + VRC01LS) | PK Step (ART + 10-1074) | Step 1 (ART + VRC01LS + 10-1074) | Step 2 (VRC01LS + 10-1074 Only) | Step 3 (ART Only)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/28 | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/28 | 1/25 | 0/28
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 23/28 | 18/25 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PK Step (ART + VRC01LS) (N=6) | PK Step (ART + 10-1074) (N=6) | Step 1 (ART + VRC01LS + 10-1074) (N=28) | Step 2 (VRC01LS + 10-1074 Only) (N=25) | Step 3 (ART Only) (N=28)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PK Step (ART + VRC01LS) (N=6) | PK Step (ART + 10-1074) (N=6) | Step 1 (ART + VRC01LS + 10-1074) (N=28) | Step 2 (VRC01LS + 10-1074 Only) (N=25) | Step 3 (ART Only) (N=28)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Eye discharge (Eye disorders) | 1 | 0 | 1 | 1 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 1 | 6 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 1 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 3
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 3 | 2 | 3 | 2
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Tinea capitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0
Tinea manuum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 5 | 8 | 7
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Buttock injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 2 | 0 | 2
Blood glucose decreased (Investigations) | 0 | 2 | 5 | 5 | 1
Blood glucose increased (Investigations) | 1 | 1 | 2 | 1 | 2
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 2 | 3 | 5 | 2
Carbon dioxide decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 4 | 2 | 8 | 7 | 14
Neutrophil count decreased (Investigations) | 1 | 1 | 10 | 4 | 8
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 7 | 11 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5 | 7 | 8
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03707977/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03707977/SAP_001.pdf
  • Informed Consent Form: PK Step (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03707977/ICF_002.pdf
  • Informed Consent Form: Steps 1 to 3 (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03707977/ICF_003.pdf